CLINICAL TRIAL: NCT02253836
Title: A Single-Centre Open-Label Study in Healthy Adult Volunteers to Assess the Pharmacokinetic Interactions Between Steady-State TPV (500 mg) and Single-Dose and Steady-State Atazanavir (300 mg QD) in the Presence of Ritonavir (100 mg)
Brief Title: Pharmacokinetic Study in Healthy Adult Volunteers to Assess the Interactions Between Steady-State Tipranavir and Atazanavir in the Presence of Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1182.61
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Atazanavir Sulfate

ARMS (1):
- TAZ/RTV - TPV/RTV - TPV/RTV+TAZ (Experimental): Days 1-9: single dose TAZ/RTV
  Days 16-23: morning and evening dose TPV/RTV
  Days 24-32: TPV/RTV + TAZ
  Interventions: Drug: Tipranavir; Drug: Ritonavir; Drug: Atazanavir

INTERVENTIONS:
Drug: Tipranavir — TPV
Drug: Ritonavir — RTV
Drug: Atazanavir — TAZ

SUMMARY:
Study to investigate the effects of steady-state TPV/r (500 mg/100 mg BID) on the single-dose and steady-state pharmacokinetics of Atazanavir (300 mg QD) co-administered with Ritonavir (100 mg). To investigate the effects of single-dose and steady-state Atazanavir (300 mg) on the steady-state pharmacokinetics of Tipranavir and Ritonavir.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 60 years of age inclusive
2. A Body Mass Index (BMI) between 18 and 29 kg/m2
3. Signed informed consent prior to trial participation
4. Ability to swallow multiple large capsules without difficulty
5. Acceptable laboratory values that indicate adequate baseline organ function at screening visit:

   * Laboratory values are considered to be acceptable if the severity of any parameter is ≤ Grade 1, based on the Division of AIDS/AIDS Clinical Trials Group Grading Scale
   * All abnormal laboratory values > Grade 1 are subject to approval by the trial clinical monitor
6. Acceptable medical history, physical examination, and 12-lead ECG at screening
7. Willingness to abstain from the following starting 2 weeks prior to administration of any study medication and up until the end of the study:

   - Grapefruit or grapefruit juice, Red wine, Seville oranges, St. John's Wort, and Milk Thistle
8. Willingness to abstain from alcohol starting 3 days prior to administration of any study medication up to the end of the study
9. Willingness to abstain from the following starting 3 days prior to pharmacokinetic (PK) sampling:

   - Garlic supplements and Methylxanthine containing foods or drinks (including coffee, tea, cola, energy drinks, chocolate, etc.)
10. Willingness to abstain from over-the-counter herbal medications for the duration of the study
11. Must be a non-smoker
12. Willingness to abstain from vigorous physical exercise during intensive PK Days 1, 9, 23, 24 and 32
13. Reasonable probability for completion of the study

Exclusion Criteria:

1. Female subjects of reproductive potential who:

   * Have positive serum pregnancy test
   * Have not been using a barrier method of contraception for at least 3 months prior to participation in the study
   * Are not willing to use a reliable method of barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam), during and 60 days after completion/termination of the trial
   * Are breast-feeding
2. Participation in another trial with an investigational medicine within 2 months prior to Day 0 of this study
3. Use of any medication listed in the protocol within 30 days prior to Day 0 of this study
4. Use of any pharmacological contraceptive (including oral, patch or injectable contraceptives) within 1 month prior to Day 0 and for the duration of the study. Due to long half-life,subjects using of Depo-Provera within six months prior to Day 0 will be excluded from participation in this study
5. Use of hormone replacement therapy within 1 month prior to Day 0 and anytime during the study
6. Administration of antibiotics within 15 days prior to Day 0 and anytime during the study
7. History of acute illness within 60 days prior to Day 0

   o Subjects will be excluded for acute illnesses that occurred more than 60 days prior to Day 0 if, in the opinion of the investigator, the subject does not qualify as a healthy volunteer
8. Have serological evidence of hepatitis B or C virus
9. Have serological evidence of exposure to HIV
10. Alcohol or substance abuse within 1 year prior to screening or during the study
11. Blood or plasma donations within 30 days prior to Day 0 or during the study
12. Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering Tipranavir, Ritonavir or Atazanavir to the subject
13. Subjects with pre-existing heart conduction abnormalities
14. Subjects who have taken (within 7 days prior to Day 0) any over-the-counter or prescription medication that, in the opinion of the investigator in consultation with the clinical monitor, might interfere with absorption, distribution, or metabolism of the study medications
15. Known hypersensitivity to sulphonamide class of drugs
16. Inability to adhere to the protocol
17. Cautions or warnings in the Ritonavir and Atazanavir package insert which, in the opinion of the investigator, constitute grounds for subject exclusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-01; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration | up to day 33
Drug concentration in plasma at 12 hr after administration for Tipranavir (TPV) and Ritonavir (RTV) | 12 hours after drug administration
Drug concentration in plasma at 24 hr after administration for Atazanavir (TAZ) | 24 hours after drug administration
Area under plasma concentration time curve from 0-12 hours (AUC0-12h) for TPV and RTV | up to 12 hours after drug administration
AUC0-24h for TAZ | up to 24 hours after drug administration

SECONDARY OUTCOMES:
Time from dosing to the maximum concentration | up to day 33
Elimination half-life | up to day 33
Oral clearance | up to day 33
Volume of distribution | up to day 33
Number of patients with adverse events | up to day 33